CLINICAL TRIAL: NCT06731660
Title: Effect of Education and Feedback, Wispr Digital Otoscope, or Both on Antibiotic Prescribing Patterns for Otitis Media in Young Children
Brief Title: Digital Otoscope Versus Education and Feedback for Otitis Media in Young Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Louis Vernacchio, Director of Research, Boston Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: P00049513
Record Dates: First submitted 2024-12-05; First posted 2024-12-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Otitis Media; Antimicrobial Stewardship
MeSH Terms: conditions — Otitis Media | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design comparing effect of Wispr digital otoscope, education with performance feedback, both, or neither on diagnosis and antibiotic treatment of otitis media in young children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Education with personalized performance feedback (Experimental): Education about proper otitis media diagnosis following criteria from the American Academy of Pediatrics with personalized performance feedback on otitis media diagnosis and treatment rates delivered via email
  Interventions: Other: Education with personalized performance feedback
- Use of digital otoscope (Experimental): Use of the Wispr digital otoscope to diagnose otitis media in place of a traditional visual otoscope
  Interventions: Device: Use of digital otoscope
- Education with personalized performance feedback plus use of a digital otoscope (Experimental): Education about proper otitis media diagnosis following criteria from the American Academy of Pediatrics with personalized performance feedback on otitis media diagnosis and treatment rates delivered via email plus use of the Wispr digital otoscope to diagnose otitis media in place of a traditional visual otoscope
  Interventions: Other: Education with personalized performance feedback; Device: Use of digital otoscope
- Control (No Intervention): Control arm, no intervention

INTERVENTIONS:
Other: Education with personalized performance feedback — Education about proper otitis media diagnosis following criteria from the American Academy of Pediatrics with personalized performance feedback on otitis media diagnosis and treatment rates delivered via email
  Other Names: Education and feedback
  Arms: Education with personalized performance feedback; Education with personalized performance feedback plus use of a digital otoscope
Device: Use of digital otoscope — Use of the Wispr digital otoscope to diagnose otitis media in place of a traditional visual otoscope
  Arms: Education with personalized performance feedback plus use of a digital otoscope; Use of digital otoscope

SUMMARY:
Randomized controlled trial involving 40 pediatric primary care clinicians with high rates of diagnosing and treating middle ear infections. Ten enrolled clinicians will be randomly assigned to each of 4 arms for a three-month trial: 1) personalized education and feedback about proper ear infection diagnosis; 2) use of a digital otoscope; 3) both education and feedback plus use of a digital otoscope; 4) control (no intervention).

DETAILED DESCRIPTION:
Randomized controlled trial involving 40 pediatric primary care clinicians with rates of otitis media diagnosis and antibiotic prescribing in the top quartile of the entire clinician population of the Pediatric Physicians' Organization at Children's over the previous 12 months who consent to enroll in the trial after direct outreach from the study team. Ten enrolled clinicians will be randomly assigned to each of 4 arms for a three-month intervention period: 1) personalized education and feedback about proper otitis media diagnosis following criteria from the American Academy of Pediatrics; 2) use of the Wispr digital otoscope; 3) both education and feedback plus use of the Wispr digital otoscope; 4) control (no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric primary care clinicians from the Pediatric Physicians' Organization at Children's with an Otitis Media Treatment Index for the previous 12 months in the top quartile of all Pediatric Physicians' Organization at Children's clinicians with at least 100 qualifying encounters in the year

Exclusion Criteria:

* Currently using any digital otoscope
* More than one other clinician from the same practice participating in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in OMTI | 3 months
  Proportion of encounters in children 6-59 months of age with any respiratory diagnosis who are diagnosed with otitis media and treated with a systemic antibiotic.

SECONDARY OUTCOMES:
Change in overall antibiotic courses prescribed | 3 months
  Courses of systemic antibiotics per 1000 children per year among children 6-59 months of age.
Change in overall prescribed antibiotic days | 3 months
  Total days of systemic antibiotics per 1000 children per year among children 6-59 months of age.
Clinician confidence and satisfaction in diagnosing OM and preference for digital versus traditional otoscope | 3 months
  Clinician responses to a pre- and post-intervention surveys regarding confidence in diagnosing otitis media and satisfaction with digital versus traditional otoscope.

OTHER OUTCOMES:
Return respiratory illness visits within 7 days (balancing measure) | 3 months
  Proportion of patients with an index encounter with respiratory diagnosis who return to the primary care office for a visit with a respiratory diagnosis within 7 days of the index visit.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Vernacchio, MD, MSc, Principal Investigator — Pediatric Physicians' Organization at Children's
Locations (1):
- Pediatric Physicians' Organization at Children's, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Electronic health record data use for the study are property of the individual practices and may not be shard publicly without their expressed permission.